CLINICAL TRIAL: NCT04704219
Title: A Phase 2, Single-arm, Open-label Clinical Trial of Pembrolizumab Plus Lenvatinib in Participants With First-line Advanced/Metastatic Non-clear Cell Renal Cell Carcinoma (nccRCC) (KEYNOTE-B61)
Brief Title: Pembrolizumab Plus Lenvatinib for First-line Advanced/Metastatic Non-clear Cell Renal Cell Carcinoma (1L nccRCC) (MK-3475-B61)
Acronym: KEYNOTE-B61
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-B61; MK-3475-B61 (Other: MSD); 2023-504944-32-00 (Registry Identifier: EU CT); U1111-1290-4553 (Registry Identifier: UTN); 2020-004087-26 (EudraCT Number)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Pembrolizumab; Lenvatinib
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Lenvatinib (Experimental): Pembrolizumab 400 mg, every 6 weeks (Q6W) intravenous (IV) up to 18 infusions or up to progressive disease or discontinuation PLUS Lenvatinib 20 mg, daily (QD), oral, until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab 400 mg, every 6 weeks (Q6W) intravenous (IV) up to 18 infusions or up to progressive disease or discontinuation.
  Other Names: KEYTRUDA®; MK-3475
Drug: Lenvatinib — Lenvatinib 20 mg, daily (QD), oral, until progressive disease or discontinuation.
  Other Names: LENVIMA®; Kisplyx; MK-7902; E7080

SUMMARY:
This study is being performed as a single-arm open-label study in order to rapidly provide information on the potential benefits of the combination of pembrolizumab and lenvatinib in participants with previously untreated advanced/metastatic non-clear cell renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a histologically confirmed diagnosis of nccRCC.
2. Has locally advanced/metastatic disease (ie, Stage IV per the American Joint Committee on Cancer).
3. Has received no prior systemic therapy for advanced nccRCC. Note: Prior neoadjuvant/adjuvant therapy for nccRCC is acceptable if completed >12 months prior to allocation.
4. Male participants agree to use approved contraception during the treatment period for at least 7 days after the last dose of study medication, or refrain from heterosexual intercourse during this period.
5. Female participants are not pregnant or breastfeeding, and are not a woman of childbearing potential (WOCBP), OR are a WOCBP that agrees to use contraception during the treatment period and for at least 120 days post pembrolizumab, or 30 days post lenvatinib, whichever occurs last.
6. Has measurable disease per RECIST 1.1 as assessed by BICR. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Has submitted an archival tumor tissue sample or newly obtained core or incisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
8. Has Karnofsky Performance Status (KPS) ≥70% as assessed within 10 days prior to the start of study intervention.
9. Has adequately controlled blood pressure with or without antihypertensive medications
10. Have adequate organ function.

Exclusion Criteria:

1. Has collecting duct histology.
2. A WOCBP who has a positive urine pregnancy test within 24 hours before the first dose of study intervention.
3. Has a left ventricular ejection fraction below the institutional (or local laboratory) normal range.
4. Has radiographic encasement or invasion of a major blood vessel, or of intratumoral cavitation.
5. Has clinically significant cardiovascular disease within 12 months from first dose of study intervention.
6. Has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
7. Has active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
8. Has had major surgery within 3 weeks prior to first dose of study intervention.
9. Has received prior therapy with an anti-programmed cell-death 1 (PD-1), anti-programmed cell-death ligand 1 (PD-L1), or anti-programmed cell-death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
10. Has received prior systemic anticancer therapy including investigational agents within 4 weeks prior to allocation.
11. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
12. Has received a live or attenuated vaccine within 30 days before the first dose of study intervention.
13. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
14. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
15. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
16. Has known active CNS metastases and/or carcinomatous meningitis.
17. Has severe hypersensitivity (≥Grade 3) to pembrolizumab, lenvatinib and/or any of their excipients.
18. Has an active autoimmune disease that has required systemic treatment in past 2 years
19. Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
20. Has an active infection requiring systemic therapy.
21. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
22. Has a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus.
23. Has a known history of active tuberculosis (TB; Bacillus tuberculosis).
24. Has had an allogenic tissue/solid organ transplant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (56):
- United States (8):
  - Georgetown University Medical Center ( Site 0001), Washington D.C., District of Columbia
  - St. Vincent Frontier Cancer Center ( Site 0004), Billings, Montana
  - Comprehensive Cancer Centers of Nevada ( Site 0010), Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center ( Site 0015), New York, New York
  - Fox Chase Cancer Center ( Site 0011), Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center ( Site 0008), Nashville, Tennessee
  - Seattle Cancer Care Alliance ( Site 0014), Seattle, Washington
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0006), Milwaukee, Wisconsin
- Australia (6):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 0405), Macquarie Park, New South Wales
  - Calvary Mater Newcastle ( Site 0403), Waratah, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Si, Brisbane, Queensland
  - Ashford Cancer Centre Research ( Site 0404), Kurralta Park, South Australia
  - Monash Health ( Site 0400), Clayton, Victoria
  - Fiona Stanley Hospital ( Site 0402), Murdoch, Western Australia
- Canada (4):
  - BC Cancer Vancouver-Clinical Trials Unit ( Site 1500), Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre ( Site 1501), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 1504), Toronto, Ontario
  - CHU de Quebec - Université Laval - Hotel Dieu de Quebec ( Site 1502), Québec, Quebec
- France (5):
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 1007), Strasbourg, Alsace
  - Centre François Baclesse ( Site 1000), Caen, Calvados
  - Centre de Cancérologie du Grand Montpellier ( Site 1005), Montpellier, Languedoc-Roussillon
  - centre hospitalier lyon sud ( Site 1003), Pierre-Bénite, Rhone
  - Gustave Roussy ( Site 1002), Villejuif, Val-de-Marne
- Hungary (4):
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Okta-Klinikai Onkológiai és Sugárterápiás C, Miskolc, Borsod-Abauj Zemplen county
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 0303), Szolnok, Jász-Nagykun-Szolnok
  - Országos Onkológiai Intézet-Urogenital Tumors Department and Clinical Pharmacology ( Site 0304), Budapest, Pest County
  - Debreceni Egyetem Klinikai Kozpont-Onkológiai Klinika ( Site 0300), Debrecen
- Tallaght University Hospital ( Site 1600), Dublin, Ireland
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli-Medical Oncology ( Site 0901), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 0903), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma-Oncology Unit ( Site 0902), Verona, Veneto
  - Azienda Ospedaliera Santa Maria Terni-SC Oncologia ( Site 0900), Terni
- Poland (3):
  - Szpital Kliniczny im. Przemienienia Panskiego Uniwersytetu M-chemotherapy department ( Site 0800), Poznan, Greater Poland Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 0802), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
- Russia (4):
  - Russian Scientific Center of Radiology-Russian Scientific Center of Radiology ( Site 0602), Moscow, Moscow
  - Volga District Medical Center-Urology Department ( Site 0604), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Nizhegorodsky Regional Oncology Dispensary, Branch #2-chemotherapy ( Site 0605), Nizhny Novgorod, Nizhny Novgorod Oblast
  - SHBI Leningrad Regional Clinical Oncology Dispensary-Clinical Trials Department ( Site 0607), Saint Petersburg
- South Korea (3):
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1302), Seoul
  - Asan Medical Center-Department of Oncology ( Site 1300), Seoul
  - Samsung Medical Center ( Site 1301), Seoul
- Spain (3):
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 0200), Madrid, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 0202), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 0201), Barcelona
- Turkey (Türkiye) (5):
  - Istanbul Universitesi Cerrahpasa ( Site 1104), Istanbul- Fatih, Istanbul
  - Ege University Medicine of Faculty ( Site 1102), Bornova, İzmir
  - Ankara University Hospital Cebeci ( Site 1105), Ankara
  - Hacettepe Universitesi-oncology hospital ( Site 1101), Ankara
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 1103), Istanbul
- Ukraine (4):
  - Cherkasy Regional Oncology Dispensary ( Site 0504), Cherkassy, Cherkasy Oblast
  - Chernihiv Medical Center of Modern Oncology ( Site 0509), Chernihiv, Chernihiv Oblast
  - Dnepropetrovsk Regional Clinical Hospital Mechnikov-Department of urology ( Site 0508), Dnipro, Dnipropetrovsk Oblast
  - CNPE "Regional Center of Oncology"-oncourology department ( Site 0502), Kharkiv, Kharkivs’ka Oblast’
- United Kingdom (2):
  - Cambridge University Hospital ( Site 1200), Cambridge, England
  - The Christie ( Site 1205), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Albiges L, Gurney H, Atduev V, Suarez C, Climent MA, Pook D, Tomczak P, Barthelemy P, Lee JL, Stus V, Ferguson T, Wiechno P, Gokmen E, Lacombe L, Gedye C, Perini RF, Sharma M, Peng X, Lee CH. Pembrolizumab plus lenvatinib as first-line therapy for advanced non-clear-cell renal cell carcinoma (KEYNOTE-B61): a single-arm, multicentre, phase 2 trial. Lancet Oncol. 2023 Aug;24(8):881-891. doi: 10.1016/S1470-2045(23)00276-0. Epub 2023 Jul 11. PMID 37451291
- [Result] Voss MH, Gurney H, Atduev V, Suarez C, Climent MA, Pook D, Tomczak P, Barthelemy P, Lee JL, Nalbandian T, Stus V, Ferguson T, Wiechno P, Gokmen E, Lacombe L, Gedye C, Cornell J, Sharma M, Burgents JE, Albiges L. First-line Pembrolizumab Plus Lenvatinib for Advanced Non-clear-cell Renal Cell Carcinoma: Updated Results from the Phase 2 KEYNOTE-B61 Trial. Eur Urol. 2025 Dec;88(6):614-624. doi: 10.1016/j.eururo.2025.05.019. Epub 2025 Jul 24. PMID 40707309
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26333&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 56 centers in 14 countries.
Pre-assignment Details: Per protocol, six participants who experienced progression of Renal Cell Carcinoma (RCC) by radiographic evaluation continued second course treatment.
Groups:
- Pembrolizumab + Lenvatinib: Participants with non-clear cell Renal Cell Carcinoma (nccRCC) received 400 mg Pembrolizumab (Pembro) intravenously (IV) on Day 1 of a 42-day cycle (every 6 weeks (Q6W)) for approximately 2 years PLUS 20 mg Lenvatinib (Lenva) orally once daily (QD) on Days 1 and 22 of a 42-day cycle (Q6W). Participants continued study intervention until progressive disease or discontinuation.
Period: Overall Study
Arm/Group | Pembrolizumab + Lenvatinib
Started | 160
Treated | 158
Second Course Treatment | 6
Completed | 0
Not Completed | 160
Not completed — Screen Failure | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 78
Not completed — Participants Ongoing | 80

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 137
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a best overall response of either Complete Response (CR): Disappearance of all target lesions or Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions as assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experienced a CR or PR as assessed per RECIST 1.1 by blinded independent central review (BICR) is presented.
Time Frame: Up to approximately 47 months
Population: All allocated participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 158
Percentage of participants | 50.6 [42.6 to 58.7]

2. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), DOR was defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. Duration of response per RECIST 1.1 by Blinded Independent Central Review (BICR) is presented.
Time Frame: Up to approximately 47 months
Population: All allocated participants who received at least 1 dose of study intervention and had confirmed complete response or partial response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 80
Months | 23.5 [16.5 to 29.5]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from date of study treatment to the first documented progressive disease (PD) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The percentage of participants who experienced PFS per RECIST 1.1 by Blinded Independent Central Review (BICR) is presented.
Time Frame: Up to approximately 47 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 158
Months | 17.9 [15.0 to 21.1]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of study treatment to the date of death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. The OS for all participants is presented.
Time Frame: Up to approximately 47 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 158
Months | 41.5 [32.8 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants who have achieved Complete Response (CR): Disappearance of all target lesions or Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm]) of ≥6 months per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR).
Time Frame: Up to approximately 47 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 158
Percentage of participants | 71.5 [63.8 to 78.4]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm]). The appearance of one or more new lesions is also considered PD]). Disease Control rate per RECIST 1.1 by Blinded Independent Central Review (BICR) is presented.
Time Frame: Up to approximately 47 months
Population: All allocated participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 158
Percentage of Participants | 82.3 [75.4 to 87.9]

7. Secondary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with at least one or more AE is presented.
Time Frame: Up to approximately 56 months
Reporting Status: Not Posted

8. Secondary Outcome: Number of Participants Who Discontinued From Study Treatment Due to an AE
Description: as for outcome 7
Time Frame: Up to approximately 56 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 56 months
Description: All-Cause Mortality included all randomized participants. Serious and Other adverse events (AEs) included all allocated participants who received at least one dose of study intervention. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study intervention. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study intervention were excluded.
Groups:
- Pembrolizumab + Lenvatinib Second Course: Participants who experienced progression of Renal Cell Carcinoma (RCC) by radiographic evaluation continued second course treatment of 400 mg Pembrolizumab (Pembro) intravenously (IV) on Day 1 of a 42-day cycle (every 6 weeks (Q6W)) for approximately 1 year PLUS 20 mg Lenvatinib (Lenva) orally once daily (QD) on Days 1 and 22 of a 42-day cycle (Q6W). Participants continued study intervention until progressive disease or discontinuation.
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Lenvatinib Second Course
All-Cause Mortality (participants affected / at risk) | 79/160 | 0/6
Serious Adverse Events (participants affected / at risk) | 76/158 | 2/6
Other Adverse Events (participants affected / at risk) | 155/158 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib (N=158) | Pembrolizumab + Lenvatinib Second Course (N=6)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure with reduced ejection fraction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Immune-mediated hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 4 (4) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib (N=158) | Pembrolizumab + Lenvatinib Second Course (N=6)
Anaemia (Blood and lymphatic system disorders) | 18 (25) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 24 (27) | 0 (0)
Hypothyroidism (Endocrine disorders) | 70 (102) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 25 (33) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 16 (21) | 0 (0)
Constipation (Gastrointestinal disorders) | 31 (39) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 88 (238) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 21 (21) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (17) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 10 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 51 (79) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 9 (10) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 33 (49) | 0 (0)
Toothache (Gastrointestinal disorders) | 8 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 27 (42) | 0 (0)
Asthenia (General disorders) | 41 (52) | 0 (0)
Chest pain (General disorders) | 11 (12) | 0 (0)
Fatigue (General disorders) | 59 (75) | 0 (0)
Mucosal inflammation (General disorders) | 25 (39) | 0 (0)
Oedema peripheral (General disorders) | 19 (22) | 0 (0)
Pyrexia (General disorders) | 14 (14) | 0 (0)
COVID-19 (Infections and infestations) | 39 (44) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 14 (26) | 0 (0)
Urinary tract infection (Infections and infestations) | 15 (27) | 0 (0)
Alanine aminotransferase increased (Investigations) | 28 (39) | 0 (0)
Amylase increased (Investigations) | 14 (35) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 29 (41) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 12 (18) | 0 (0)
Blood bilirubin increased (Investigations) | 8 (12) | 0 (0)
Blood creatinine increased (Investigations) | 20 (31) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 18 (19) | 0 (0)
Lipase increased (Investigations) | 17 (25) | 0 (0)
Weight decreased (Investigations) | 46 (58) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 54 (72) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (8) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 15 (16) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (14) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 (90) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (10) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (31) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 23 (29) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (17) | 0 (0)
Dizziness (Nervous system disorders) | 17 (17) | 0 (0)
Dysgeusia (Nervous system disorders) | 17 (20) | 0 (0)
Headache (Nervous system disorders) | 36 (45) | 0 (0)
Insomnia (Psychiatric disorders) | 15 (17) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 10 (11) | 0 (0)
Proteinuria (Renal and urinary disorders) | 59 (93) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (37) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 51 (67) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (14) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 50 (84) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (40) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 23 (24) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (20) | 0 (0)
Hypertension (Vascular disorders) | 95 (174) | 0 (0)
Hypotension (Vascular disorders) | 8 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity was not directed by the Sponsor, the investigator agreed to submit all manuscripts or abstracts to the Sponsor before submission. This allowed the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT04704219/Prot_SAP_000.pdf